CLINICAL TRIAL: NCT03268291
Title: Impact of Communicational Program "Trust" on Adherence to Medications in Patients With Prior Myocardial Infarction Who Underwent Successful Revascularization by Stenting or Thrombolysis: A Prospective Multicenter Randomized Trial
Brief Title: Communicational Program "Trust" to Improve Adherence to Medications
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Call of Trust
Record Dates: First submitted 2017-08-29; First posted 2017-08-31 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Coronary Artery Disease; Myocardial Infarction; Cardiovascular Diseases
Keywords: Adherence to therapy; Myocardial Infarction; Coronary Artery Disease; Communicational program
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: The study will include 2,000 patients. Patients will be randomized into two groups: standard outpatient observation (n = 1 000), the "Trust" program (n = 1 000).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard outpatient observation (Active Comparator): Outpatient management according to Ministry of health standards
  Interventions: Other: Standard outpatient observation
- Communicational program "Trust" (Experimental): The developed program is based on the experience of international research studies and includes the following sections:
  * daily seminars with patients going to be discharged about the benefits of adherence to therapy; distribution of printed materials;
  * service for the regular informing of the patients which is motivating to remain adherence to medications by automated contact management systems (SMS, e-mail), as well as calls from contact center operators;
  * questioning of participants of the program for general adherence to therapy, reasons for refusal, change of therapy / drug, complaints and other. The questioning is carried out through telephone interviewing by contact center operators and automatic collection of electronic forms through aggregator services.
  Interventions: Behavioral: Communicational program "Trust"

INTERVENTIONS:
Other: Standard outpatient observation — Outpatient management according to Ministry of health standards
  Arms: Standard outpatient observation
Behavioral: Communicational program "Trust" — The developed program is based on the experience of international research studies and includes the following sections:
  daily seminars with patients going to be discharged about the benefits of adherence to therapy; distribution of printed materials; service for the regular informing of the patients which is motivating to remain adherence to medications by automated contact management systems (SMS, e-mail), as well as calls from contact center operators; questioning of participants of the program for general adherence to therapy, reasons for refusal, change of therapy / drug, complaints and other. The questioning is carried out through telephone interviewing by contact center operators and automatic collection of electronic forms through aggregator services.
  Arms: Communicational program "Trust"

SUMMARY:
The trial was designed in such a way as to show that the proposed program "Trust" increases the proportion of patients who adhere to therapy in the cohort of those with coronary heart disease for two years after successful revascularization by using thrombolytic or stenting of the coronary arteries against the background of myocardial infarction.

DETAILED DESCRIPTION:
The "Trust" program includes a set of measures aimed at increasing the level of adherence to therapy in patients with myocardial infarction. Differences in adherence rates between patients enrolled in the program and patients undergoing standard outpatient care will be monitored during the study. The study will be conducted according to the clinical approbation protocol, the principles of good clinical practice (GCP) and regulatory requirements.

The developed program is based on the experience of international research studies and includes the following sections:

* daily seminars with patients going to be discharged about the benefits of adherence to therapy; distribution of printed materials;
* service for the regular informing of the patients which is motivating to remain adherence to medications by automated contact management systems (SMS, e-mail), as well as calls from contact center operators;
* questioning of participants of the program for general adherence to therapy, reasons for refusal, change of therapy / drug, complaints and other. The questioning is carried out through telephone interviewing by contact center operators and automatic collection of electronic forms through aggregator services.

Information motivating to remain adherence to the therapy is structured as follows:

A) greeting and presentation, a reminder of the necessity for therapy, with the support of the patient's Trust in prolonging the quality of life by regular use of medications; B) the explanation of the action of the medicine taking into account the peculiarities of ordinary consciousness, warning the patient of the most common mistakes in treatment; C) recommendations for changing lifestyle and explaining their need; D) a reminder of the possibility to contact the attending physician, emotional support and counseling.

The establishment of an information and counseling center will allow the patient to be supported throughout the time when the likelihood of giving up therapy and the risk of complications due to failure are most likely.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Recent acute myocardial infarction within the past 2 months
* Successful revascularization via coronary stenting or thrombolysis

Exclusion Criteria:

* Concomitant cardiovascular disorders requiring surgical treatment
* Coronary revascularization via CABG
* Patient refused from participating
* Patient is not available for communication within 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Medication Adherence | During 1 year
  Adherence to every class of prescribed medications: Acetylsalicylic acid, P2Y12 receptor inhibitors, Beta-blockers, ACE inhibitors according to percent of medication taking days. Adherence above 80% will be satisfactory

CONTACTS AND LOCATIONS:
Locations (1):
- State Research Institute of CIrculation Pathology, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: Yes
All the data
Supporting Information: Study Protocol, CSR